CLINICAL TRIAL: NCT00088933
Title: Randomized Single Institution Pilot Study of Vaccinia-CEA(6D)-TRICOM and Fowlpox-CEA(6D)-TRICOM With GM-CSF in Combination With Docetaxel in Patients With CEA-Bearing Cancers
Brief Title: Vaccine Therapy and Sargramostim With or Without Docetaxel in Treating Patients With Metastatic Lung Cancer or Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00049; NCI-2009-00049 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000377574; 02-452; 02-452 (Other: Lombardi Comprehensive Cancer Center at Georgetown University); 6230 (Other: CTEP); R01CA088972 (NIH); P30CA051008 (NIH)
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2013-03

CONDITIONS: Extensive Stage Small Cell Lung Cancer; Recurrent Colon Cancer; Recurrent Non-small Cell Lung Cancer; Recurrent Rectal Cancer; Recurrent Small Cell Lung Cancer; Stage IV Colon Cancer; Stage IV Non-small Cell Lung Cancer; Stage IV Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Carcinoma, Non-Small-Cell Lung; Rectal Neoplasms; Small Cell Lung Carcinoma | interventions — Docetaxel; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor

ARMS (6):
- Arm I (Experimental): Three weeks after treatment with vaccinia-CEA-TRICOM vaccine, patients receive fowlpox-CEA-TRICOM vaccine SC on day 1 and GM-CSF SC into each vaccination site on days 1-4.
  Interventions: Drug: recombinant fowlpox-CEA(6D)/TRICOM vaccine; Drug: recombinant vaccinia-CEA(6D)-TRICOM vaccine; Drug: sargramostim
- Arm II (Experimental): Patients receive fowlpox-CEA-TRICOM vaccine and GM-CSF as in arm I and lower-dose docetaxel IV over 30 minutes on days 1 and 8.
  Interventions: Drug: recombinant fowlpox-CEA(6D)/TRICOM vaccine; Drug: recombinant vaccinia-CEA(6D)-TRICOM vaccine; Drug: docetaxel; Drug: sargramostim
- Arm III (Experimental): Patients receive fowlpox-CEA-TRICOM vaccine and GM-CSF as in arm I and standard-dose docetaxel IV over 30 minutes on days 1 and 8.
  Interventions: Drug: recombinant fowlpox-CEA(6D)/TRICOM vaccine; Drug: recombinant vaccinia-CEA(6D)-TRICOM vaccine; Drug: docetaxel; Drug: sargramostim
- Arm IV (Experimental): Patients receive fowlpox-CEA-TRICOM vaccine and GM-CSF as in arm I and full-dose docetaxel IV over 1 hour on day 1.
  Interventions: Drug: recombinant fowlpox-CEA(6D)/TRICOM vaccine; Drug: recombinant vaccinia-CEA(6D)-TRICOM vaccine; Drug: docetaxel; Drug: sargramostim
- Arm V (Experimental): Patients receive full-dose docetaxel IV over 1 hour on day 1, fowlpox-CEA-TRICOM vaccine SC on day 8, and GM-CSF SC into each vaccination site on days 8-11.
  Interventions: Drug: recombinant fowlpox-CEA(6D)/TRICOM vaccine; Drug: recombinant vaccinia-CEA(6D)-TRICOM vaccine; Drug: docetaxel; Drug: sargramostim
- Arm VI (Experimental): Patients receive full-dose docetaxel as in arm V, fowlpox-CEA-TRICOM vaccine SC on day 15, and GM-CSF SC into each vaccination site on days 15-18.
  Interventions: Drug: recombinant fowlpox-CEA(6D)/TRICOM vaccine; Drug: recombinant vaccinia-CEA(6D)-TRICOM vaccine; Drug: docetaxel; Drug: sargramostim

INTERVENTIONS:
Drug: recombinant fowlpox-CEA(6D)/TRICOM vaccine — Given intradermally
  Other Names: fowlpox-CEA-B7-1/ICAM-1/LFA-3; rF-CEA(6D)TRICOM
Drug: recombinant vaccinia-CEA(6D)-TRICOM vaccine — Given intradermally
  Other Names: rV-CEA(6D)-TRICOM
Drug: docetaxel — Given IV
  Other Names: RP 56976; Taxotere; TXT
  Arms: Arm II; Arm III; Arm IV; Arm V; Arm VI
Drug: sargramostim — Given subcutaneously
  Other Names: GM-CSF; Leukine; Prokine

SUMMARY:
This randomized phase I trial studies the side effects, best way to give, and best dose of docetaxel when given together with vaccine therapy and sargramostim in treating patients with metastatic lung cancer or metastatic colorectal cancer. Vaccines may make the body build an immune response to kill tumor cells. Colony-stimulating factors such as sargramostim increase the number of immune cells found in bone marrow and peripheral blood. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining vaccine therapy and sargramostim with docetaxel may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the recommended dose and schedule of docetaxel when given in combination with recombinant vaccinia-CEA-TRICOM vaccine, recombinant fowlpox-CEA-TRICOM vaccine, and sargramostim (GM-CSF), defined by best immune response with acceptable toxicity, in patients with carcinoembryonic antigen (CEA)-expressing metastatic lung or colorectal cancer.

II. Compare the effect of varying doses and schedules of docetaxel on CEA-specific T-cell immune responses by ELISPOT assay in patients treated with these regimens.

III. Compare objective antitumor response in patients treated with these regimens.

OUTLINE:

This is a 2-part, randomized, pilot study. Patients are randomized to 1 of 6 treatment arms: arms I, II, and III in part I (lung cancer and colorectal cancer patients) and arms IV, V, and VI in part II (lung cancer patients only). Patients are stratified according to disease site and HLA-A2 positivity (positive vs negative). At least 6 of 10 patients must be HLA-A2 positive for each of the treatment arms.

Vaccinia-CEA-TRICOM vaccine (parts I and II): In all treatment arms, patients receive vaccinia-CEA-TRICOM vaccine intradermally on day 1 and sargramostim (GM-CSF) subcutaneously (SC) into the vaccine site on days 1-4.

Fowlpox-CEA-TRICOM vaccine and concurrent chemotherapy:

Part I (lung cancer and colorectal cancer patients):

ARM 1: Three weeks after treatment with vaccinia-CEA-TRICOM vaccine, patients receive fowlpox-CEA-TRICOM vaccine SC on day 1 and GM-CSF SC into each vaccination site on days 1-4.

ARM II: Patients receive fowlpox-CEA-TRICOM vaccine and GM-CSF as in arm I and lower-dose docetaxel IV over 30 minutes on days 1 and 8.

ARM III: Patients receive fowlpox-CEA-TRICOM vaccine and GM-CSF as in arm I and standard-dose docetaxel IV over 30 minutes on days 1 and 8.

Part II (lung cancer patients only):

ARM IV: Patients receive fowlpox-CEA-TRICOM vaccine and GM-CSF as in arm I and full-dose docetaxel IV over 1 hour on day 1.

ARM V: Patients receive full-dose docetaxel IV over 1 hour on day 1, fowlpox-CEA-TRICOM vaccine SC on day 8, and GM-CSF SC into each vaccination site on days 8-11.

ARM VI: Patients receive full-dose docetaxel as in arm V, fowlpox-CEA-TRICOM vaccine SC on day 15, and GM-CSF SC into each vaccination site on days 15-18.

Treatment in all arms repeats every 21 days for a total of 4 courses in the absence of disease progression or unacceptable toxicity. Patients who do not have significant disease progression or unacceptable toxicity after 4 courses of treatment may receive additional fowlpox-CEA-TRICOM vaccine and docetaxel according to the treatment arm on which they were enrolled at study entry. Patients are followed every 6 months for 2 years and then annually for 13 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed lung OR colorectal cancer
* Incurable metastatic disease
* Currently available standard treatment not likely to offer a survival advantage or result in superior palliation
* Evaluable disease by radiograph
* Tumor must currently express carcinoembryonic antigen (CEA) by immunohistochemistry OR CEA >= 10 ng/mL at any point during disease course
* No clinically active brain metastases
* Must have had first- and second-line treatment OR declined second-line treatment (part I only)
* Patients with colon cancer must have had or have been offered treatment with oxaliplatin (part I only)
* ECOG 0-1
* Life expectancy of at least 4 months
* Absolute neutrophil count >= 1,500/mm^3
* WBC >= 3,000/mm^3
* Platelet count >= 100,000/mm^3
* Bilirubin normal
* Meets 1 of the following criteria:

  * SGOT and SGPT =< 2.5 times upper limit of normal (ULN) AND alkaline phosphatase normal
  * SGOT and SGPT =< normal AND alkaline phosphatase =<4.0 times ULN
* Hepatitis B and C negative by clinical history and physical exam
* Creatinine =< 1.5 mg/dL OR creatinine clearance >= 60 mL/min
* Proteinuria =< grade 1
* No known or suspected history of impaired cardiac function as evidenced by baseline echocardiogram
* Adequate pulmonary function
* No history or clinical evidence of immune deficiency or autoimmunity
* HIV negative
* No history of or concurrent diagnosis of any of the following:

  * Altered immunodeficiency
  * Eczema or other eczematoid skin disorders
  * Acute, chronic, or exfoliative skin condition (e.g., atopic dermatitis, burns, impetigo, varicella zoster, severe acne, or other open rashes or wounds)
* No history of allergy or untoward reaction to prior vaccination with vaccinia virus
* No history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* No history of allergy to eggs or egg products
* No frequent vomiting or severe anorexia
* No inflammatory bowel disease
* No Crohn's disease
* No ulcerative colitis
* No active diverticulitis
* Neuropathy =< grade 1 (sensory neuropathy)
* No uncontrolled seizure disorder
* No encephalitis
* No multiple sclerosis
* Must be maintaining a reasonable state of nutrition (=< 10 % weight loss in the past month)
* Must be able to avoid close household contact (defined as sharing housing or having close physical contact) for at least 3 weeks after recombinant vaccinia vaccination with individuals with active or a history of eczema or other eczematoid skin disorders
* Must be able to avoid close household contact (defined as sharing housing or having close physical contact) for at least 3 weeks after recombinant vaccinia vaccination with those with unresolved acute, chronic, or exfoliative skin conditions (e.g., atopic dermatitis, burns, impetigo, varicella zoster, severe acne, or other open rashes or wounds)
* Must be able to avoid close household contact (defined as sharing housing or having close physical contact) for at least 3 weeks after recombinant vaccinia vaccination with any of the following individuals: pregnant or nursing women; children =< 5 years of age; immunodeficient or immunosuppressed individuals (by disease or therapy), including HIV infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 6 months after study participation
* No other concurrent serious medical illness that would preclude study participation
* No concurrent biologic therapy
* No other concurrent immunotherapy
* At least 6 weeks since prior nitrosoureas or mitomycin
* Prior docetaxel allowed (part I only)
* No prior docetaxel (part II only)
* No other concurrent chemotherapy
* No concurrent systemic steroids except for the following:

  * physiologic doses for systemic steroid replacement therapy
  * local (topical, nasal, or inhaled) steroid use
  * no concurrent steroid eye drops
  * premedication prior to and after docetaxel
* No concurrent hormonal therapy
* No prior radiotherapy to > 50 % of all nodal groups
* More than 21 days since prior major surgery
* No prior splenectomy
* Recovered from prior therapy
* At least 3-4 weeks since prior cytotoxic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-06; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Anti-tumor response rate defined as the number of patients in each arm achieving a complete or partial response or stable disease divided by the total number of patients on each arm measured according to standard RECIST guidelines | Up to 6 years
Immune response defined as the numbers of patients who achieve an ELISPOT result of 1/30,000 or higher divided by the number of HLA-A2 positive individuals for each treatment arm | Up to 6 years
  The actual ELISPOT will be recorded for each individual and will be presented graphically.
Number of patients experiencing each of the toxicities by grade for each treatment arm | Up to 6 years

SECONDARY OUTCOMES:
Average quantity of circulating CEA cells determined by quantitative real time RT-PCR | Up to 6 years
  The impact of the combination therapy on CCC will be presented graphically with descriptive statistics. Will be plotted for each time point by each treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: John Marshall, Principal Investigator — Lombardi Comprehensive Cancer Center at Georgetown University
Locations (1):
- Lombardi Comprehensive Cancer Center at Georgetown University, Washington D.C., District of Columbia, United States